CLINICAL TRIAL: NCT01226459
Title: A Phase 3 Multi-Center Parallel Design Clinical Trial to Compare the Efficacy and Safety of 5% Minoxidil Foam vs. Vehicle in Females for the Treatment of Female Pattern Hair Loss (Androgenetic Alopecia)
Brief Title: Clinical Trial in Females for Female Pattern Hair Loss
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Healthcare Products Division of McNEIL-PPC, Inc. (Industry)
Collaborators: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MINALO3005; 2010-019881-96 (EudraCT Number)
Record Dates: First submitted 2010-10-20; First posted 2010-10-22 (Estimated); Results first posted 2014-06-03 (Estimated); Last update posted 2014-06-10 (Estimated); Status verified 2014-06

CONDITIONS: Androgenetic Alopecia
Keywords: Female Pattern Baldness
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Minoxidil Foam (Experimental): 5% Minoxidil Topical Foam
  Interventions: Drug: 5% Minoxidil Topical Foam
- Vehicle Foam (Placebo Comparator): Vehicle Topical Foam
  Interventions: Drug: Vehicle Topical Foam

INTERVENTIONS:
Drug: 5% Minoxidil Topical Foam — Dosage Form: 5% Minoxidil Topical Foam applied to the scalp; Dosage: half a cap, equivalent to 1 g of foam; Frequency: once every day; Duration: 24 weeks
  Other Names: Not yet marketed
  Arms: Minoxidil Foam
Drug: Vehicle Topical Foam — Dosage Form: Vehicle Topical Foam applied to the scalp; Dosage: half a cap, equivalent to 1 g of foam; Frequency: once every day; Duration: 24 weeks
  Other Names: Vehicle Control (Placebo)
  Arms: Vehicle Foam

SUMMARY:
This is a six month clinical trial to evaluate the effectiveness and safety in women with Female Pattern Hair Loss (FPHL), comparing a 5% minoxidil topical foam (MTF) formulation applied once a day versus a topical foam vehicle (placebo) formulation applied once a day.

DETAILED DESCRIPTION:
This is a phase 3, two-arm, randomized, double-blind, vehicle-controlled, multi-center, 24-week, parallel design trial to evaluate the efficacy and safety in women with Female Pattern Hair Loss (FPHL), comparing the 5% MTF formulation versus the foam vehicle formulation.

This clinical trial is designed to compare the risk/benefit profile of the new 5% MTF formulation applied once a day (OD) versus the foam vehicle formulation applied once a day (OD), using objective efficacy measures and safety assessments.

Study centers will screen a sufficient number of participants so that a minimum of 300 female participants with FPHL will be enrolled, to ensure 260 complete. There will be at least 16 participants enrolled per center at multiple centers located across the US and globally. Approximately 300 participants will be randomly assigned in a 1:1 ratio to use either 5% MTF OD or foam vehicle OD, for 24 weeks for efficacy and safety evaluations.

Participants meeting the inclusion criteria will be randomly assigned in the order of their enrollment at each site. The signing of the informed consent and assignment of a participant number to a subject shall constitute enrollment.

During the trial following enrollment at Baseline, participants will return to the study site at Weeks 1, 6, 12, 18 and 24 for safety assessments, adverse events monitoring, and compliance assessments. At the Week 12 and 24 visits, efficacy assessments will also be conducted, using Target Area Hair Counts (TAHC), measured by macrophotography.

ELIGIBILITY:
Inclusion Criteria:

* females, age 18 or older in general good health
* exhibits female pattern hair loss
* signs and dates an informed consent document
* agrees to use an adequate method of birth control; if of childbearing potential
* shows a negative urine pregnancy test at Screening Visit
* is willing to maintain the same hair style, hair color, and hair regimen throughout the study
* is willing and able to comply with scheduled visits, treatment plan, laboratory tests and other trial procedures

Exclusion Criteria:

* hypersensitivity to the (study product), or any ingredients of the (study product)
* known allergy to hair dye, or hair dye components
* clinically relevant history of hypotension
* untreated or uncontrolled hypertension
* pregnant, planning a pregnancy or nursing a child
* history of hair transplants
* currently use hair weaves or non-breathable wigs
* dermatologic disorders of the scalp that require chronic use of medication for control
* other types or history of hair loss
* enrolled in any other investigational medication (drug) study currently, or within the last 6 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 404 (Actual)
Dates: Start 2010-09; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clare Kendall, Study Director — Johnson & Johnson Consumer and Personal Products Worldwide
Locations (16):
- United States (12):
  - Axis Clinical Trials, Los Angeles, California
  - Therapeutics Clinical Research, San Diego, California
  - Heartland Research Associates LLC, Wichita, Kansas
  - Callender Skin & Laser Center, Glenn Dale, Maryland
  - Michigan Center for Skin Care Research, Clinton Township, Michigan
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - New York University School of Medicine, New York, New York
  - Derm Research Center of New York, Stony Brook, New York
  - Cleveland Clinic, Cleveland, Ohio
  - J&S Studies, Inc., College Station, Texas
  - David A. Whiting, MD PA, Dallas, Texas
  - The Education & Research Foundation Inc, Lynchburg, Virginia
- Hôpital Saint Jacques Service de Dermatologie, Besançon, France
- Germany (2):
  - Clinical Research Center for Hair and Skin Science Universitätsmedizin Berlin, Berlin
  - Dermaticum Practice for Dermatology, Freiburg im Breisgau
- George Eliot Hospital, Nuneaton, United Kingdom

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vehicle Foam | Minoxidil Foam
Started | 201 | 203
Completed | 180 | 171
Not Completed | 21 | 32
Not completed — Adverse Event | 2 | 8
Not completed — Protocol Violation | 4 | 3
Not completed — Withdrawal by Subject | 10 | 13
Not completed — Lost to Follow-up | 4 | 8
Not completed — Pregnancy | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent to Treat (ITT) population defined as all participants randomly assigned to a treatment group who received dispensed investigational product.
Groups:
- Total: Total of all reporting groups
Arm/Group | Vehicle Foam | Minoxidil Foam | Total
Number analyzed (Participants) | 201 | 203 | 404
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 148 | 157 | 305
  >=65 years | 53 | 46 | 99
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 201 | 203 | 404
  Male | 0 | 0 | 0
Race (NIH/OMB) [Number; unit: participants] — One participant in minoxidil foam group had no information on race and hair loss duration
  participants
    American Indian or Alaska Native | 3 | 1 | 4
    Asian | 3 | 4 | 7
    Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
    Black or African American | 55 | 50 | 105
    White | 140 | 145 | 285
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Target Area Hair Count
Description: Number of hairs in the area being examined as measured by macrophotography.
Time Frame: Baseline to Week 24
Population: Intent to Treat (ITT) population defined as all participants randomly assigned to a treatment group who received dispensed investigational product. Four participants in vehicle group and 3 participants in minoxidil foam group had no hair information at Baseline.
Measure: Mean (Standard Deviation); unit: hairs per centimeter squared
Arm/Group | Vehicle Foam | Minoxidil Foam
Number analyzed (Participants) | 197 | 200
hairs per centimeter squared
  Baseline | 152.7 (59.7) | 158.6 (61.6)
  Week 24 | 162.2 (63.1) | 175.7 (65.1)
  Change from Baseline to Week 24 | 4.0 (16.2) | 13.5 (22.3)
Statistical Analysis 1: Comparison: Vehicle Foam vs Minoxidil Foam; Intent to Treat (ITT) population defined as all participants randomly assigned to a treatment group who received dispensed investigational product. Four participants in vehicle group and 3 participants in foam group had no hair information at Baseline. Statistical analysis is of the change from baseline to week 24 data; Test type: Superiority or Other; p < 0.0001, ANCOVA; P-value is from ANCOVA model with treatment and center as factors and Baseline hair count as a covariate; Mean Difference (Final Values) = 9.1, 95% CI 2-sided [5.0 to 13.1]

2. Secondary Outcome: Target Area Hair Count
Description: Number of hairs in the area being examined as measured by macrophotography.
Time Frame: Baseline to Week 12
Population: Intent to Treat (ITT) population defined as all participants randomly assigned to a treatment group who received dispensed investigational product. Four participants in the vehicle foam group and 3 participants in the minoxidil foam group had no hair count information at Baseline.
Measure: Mean (Standard Error); unit: hairs per centimeter squared
Arm/Group | Vehicle Foam | Minoxidil Foam
Number analyzed (Participants) | 197 | 200
hairs per centimeter squared
  Baseline | 152.7 (59.7) | 158.6 (61.6)
  Week 12 | 163.3 (63.2) | 178.1 (66.4)
  Change from Baseline to Week 12 | 5.4 (15.3) | 16.4 (21.5)
Statistical Analysis 1: Comparison: Vehicle Foam vs Minoxidil Foam; Statistical analysis is of the change from baseline to week 12 data; Test type: Superiority or Other; p < 0.0001, ANCOVA; P-value is from ANCOVA model with treatment and center as factors and Baseline hair count as a covariate; Mean Difference (Final Values) = 10.8, 95% CI 2-sided [7.0 to 14.7]

3. Primary Outcome: Subject Assessment of Scalp Coverage
Description: Subject assessment of scalp coverage at Week 24 was measured as change from Baseline on a 7-point scale where 0 meant no perceived change in scalp coverage, +1 to +3 indicated progressively increased levels of scalp coverage, and -1 to -3 indicated progressively decreased levels.
Time Frame: Week 24
Population: Intent to Treat (ITT) population defined as all participants randomly assigned to a treatment group who received dispensed investigational product. Eighteen participants in vehicle foam group and 23 participants in minoxidil foam group had no scalp coverage information.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Vehicle Foam | Minoxidil Foam
Number analyzed (Participants) | 183 | 180
scores on a scale | 0.06 (1.66) | 0.74 (1.71)
Statistical Analysis 1: Comparison: Vehicle Foam vs Minoxidil Foam; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 0.69, 95% CI 2-sided [0.35 to 1.04]

ADVERSE EVENTS:
Arm/Group | Vehicle Foam | Minoxidil Foam
Serious Adverse Events (participants affected / at risk) | 4/201 | 6/203
Other Adverse Events (participants affected / at risk) | 57/201 | 63/203
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vehicle Foam (N=201) | Minoxidil Foam (N=203)
Ovarian Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine Leiomyoma (Nervous system disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 1 | 0
Cardiovascular Disorder (Cardiac disorders) | 0 | 1 — Death (1 participant died from cardiovascular disease)
Cor Pulmonale Acute (Cardiac disorders) | 1 | 0
Asthenia (General disorders) | 2 | 0
Fatigue (General disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 — Death (1 participant died from both renal failure and dehydration). Note that this is the same participant that died from renal failure.
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Memory Impairment (Nervous system disorders) | 1 | 0
Mental Status Changes (Psychiatric disorders) | 1 | 0
Post-Traumatic Stress Disorder (Psychiatric disorders) | 1 | 0
Renal Failure (Renal and urinary disorders) | 0 | 1 — Death (1 participant died from both renal failure and dehydration). Note that this is the same participant who died from dehydration.
Hypertensive Crisis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2.0% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vehicle Foam (N=201) | Minoxidil Foam (N=203)
Nasopharyngitis (Infections and infestations) | 13 | 11
Upper Respiratory Tract Infection (Infections and infestations) | 8 | 5
Sinusitis (Infections and infestations) | 5 | 7
Gastroenteritis (Infections and infestations) | 1 | 6
Urinary Tract Infection (Infections and infestations) | 1 | 4
Weight Increased (Investigations) | 14 | 17
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 5
Headache (Nervous system disorders) | 8 | 6
Hypertension (Vascular disorders) | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Multi-Center Publication will be the first publication to present the results of the Study. Upon such Multi-Center Publication, or the earlier of (a) Sponsor's confirmation that there will be no Multi-Center Publication or presentation, or (b) 12 months after the completion of the entire multi-center study, Institution and Investigator may publish or present Study data and results generated in their performance of the Study in accordance with the terms of this Article.